CLINICAL TRIAL: NCT00399737
Title: Effects of Peptides Derived From Fermented Milk on Blood Pressure Regulation System in Healthy Volunteers.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Danone Institute International (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NU167
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2006-11-15 (Estimated); Status verified 2006-11

CONDITIONS: Healthy
Keywords: ACE activity; Fermented milk peptides; Healthy male volunteers

INTERVENTIONS:
Drug: repeated intake of fermented milk followed by a single oral dose of an ACE inhibitor

SUMMARY:
Several milk proteins are precursors of peptides, released during fermentation, which possess various biochemical and physiological properties. Among them, some peptides have been reported to inhibit angiotensin-converting enzyme (ACE) in vitro (an enzyme implicated in blood pressure regulation) and to lower blood pressure (BP). in hypertensive rats and in a small sample of patients with hypertension. One possible mechanism for the BP lowering effect is inhibition of ACE. Prior investigating BP lowering effect of these peptides in a large cohort of hypertensive patients, it is necessary to assess in depth their potency to inhibit ACE in vivo in humans and to compare it to that induced by a well-known ACE inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* aged between 18 and 35 years
* informed written consent

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2005-10; Study Completion 2005-11

PRIMARY OUTCOMES:
ACE activity

SECONDARY OUTCOMES:
kinetics/dynamics

CONTACTS AND LOCATIONS:
Overall Officials: Michel Azizi, Principal Investigator — APHP
Locations (1):
- Clinical Investigation Center 920, Hôpital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Result] FitzGerald RJ, Murray BA, Walsh DJ. Hypotensive peptides from milk proteins. J Nutr. 2004 Apr;134(4):980S-8S. doi: 10.1093/jn/134.4.980S. PMID 15051858